CLINICAL TRIAL: NCT01634646
Title: A Placebo-Controlled Pilot Study to Observe the Impact Lyzme5 Has on Cholesterol and Body Weight in Man
Brief Title: Observational Study of Lyzme5 Impact on Cholesterol and Body Weight in Man
Acronym: Lyzme5
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit sufficient local qualifying volunteers for study.
Sponsor: Jeff Golini (Industry)
Collaborators: All American Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, Jeff Golini, President and Executive Scientist, All American Pharmaceutical
Organization: All American Pharmaceutical (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Double
Other Study IDs: Lyzme5-IRB26715/1
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Overweight; Elevated Cholesterol
Keywords: Observational study
MeSH Terms: conditions — Overweight; Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Overweight, elevated total cholesterol (Placebo Comparator): All individuates enrolled in this study are at least 15 lbs over their ideal weight as described on a BMI chart. Each individual must also have a total cholesterol of at least 200 mg/dl, or higher.
  Interventions: Dietary Supplement: Lyzme5

INTERVENTIONS:
Dietary Supplement: Lyzme5 — Dietary Supplement (or placebo):
  Lyzme5 (or the placebo) is to be mixed with 4 fluid ounces of a sugar free flavored drink (example: kool aid, crystal light, flavored tea drink, etc.).
  Week one:
  A single serving of the assigned material (Lyzme5 or the placebo) each day, 20 minutes before breakfast;
  Week two:
  Two (2) servings of the assigned material each day - the first, 20 minutes before breakfast and the second 20 minutes before the noon meal;
  Week three through the end of the study:
  Three (3) servings per day of the assigned material - the first, 20 minutes before breakfast, the second, 20 minutes before the noon meal, and the third, 20 minutes before the last meal of the day.

SUMMARY:
This observational placebo-controlled pilot study is intended to document whether or not Lyzme5, an over-the-counter (OTC) proprietary nutritional supplement product can positively impact, (a) weight and, (b) cholesterol levels in man.

DETAILED DESCRIPTION:
Lyzme5 is a nutritional supplement, according to the Dietary Supplement Health and Education Act (DSHEA) of 1994. It is composed of B Vitamins along with a non-essential amino acid. The individual components of this supplement are individually Generally Recognized as Safe (have GRAS status). The manufacturer's objective was to create a nutritional supplement that would have the potential to positively impact body weight, and possibly one or more lipid value (i.e., total cholesterol, LDL, triglycerides)as well, in overweight individuals who may also have minimally elevated cholesterol levels.

This observational clinical study will seek to recruit 100 volunteers in order to observe whether or not the weight-loss potential of Lyzme5, previously observed earlier in three volunteers, can be duplicated within a larger group.

The second objective is to establish whether or not Lyzme5 can positively impact cholesterol levels in man.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years of age or older;
* Able to read, understanding, and signing a consent form;
* Not pregnant or breast feeding (female only);
* Have normal bio-markers for liver and kidney function (determined by blood test);
* Being at least 15 lbs over your ideal weight as defined by the Body Mass Index [BMI] chart;
* Have a total cholesterol level of or in excess of 200 mg/dl (determined by blood test);
* Not using any illegal substances, including marijuana (medicinal or otherwise);
* Not using any "recreational drugs"
* Weighing less than 300 lbs

Exclusion Criteria:

* Under 21 years of age;
* Mentally impaired;
* Pregnant or breast feeding;
* A diabetic;
* Having digestion problems;
* Problems with kidneys, heart, or liver;
* Having, or have had cancer;
* Taking a prescription;
* Weight of 300 lbs or over;
* Total cholesterol under 200 mg/dl;
* Using "recreational" drugs.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Weight loss | 60 days post initiation
  Volunteers will be weighed at the beginning and end of their 60 day participation. Weight loss (or gain) will be assessed.

SECONDARY OUTCOMES:
Cholesterol reduction | 60 days post initiation
  The following will be assessed at enrollment, after 30 days, and at the conclusion of the volunteer's 60 day participation: Total cholesterol, HDL, LDL, and triglyceride levels.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Golini, Principal Investigator — All American Pharmaceutical
Locations (1):
- All American Pharmaceutical and Natural Foods Corporation, Billings, Montana, United States